CLINICAL TRIAL: NCT01286636
Title: Artificial Neural Network Directed Therapy of Severe Obstructive Sleep Apnea
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ali El Solh, Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ANN02
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Apnea
Keywords: artificial neural network
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- artificial neural network (Experimental)
  Interventions: Other: computer model
- Polysomnogram (Active Comparator)
  Interventions: Other: Polysomnogram

INTERVENTIONS:
Other: computer model — Diagnosis of Sleep apnea and treatment guidance will rely on a computer model prediction.
  Arms: artificial neural network
Other: Polysomnogram — Diagnosis of sleep apnea will rely on polysomnogram
  Arms: Polysomnogram

SUMMARY:
The investigators have developed a simple, accurate, and a point-of-care, computer-based clinical decision support system (CDSS) not only to detect the presence of sleep apnea but also to predict its severity. The CDSS is based on deploying an artificial neural network (ANN) derived from anthropomorphic and clinical characteristics.

The investigators hypothesize that patients with severe OSA defined as AHI≥30 can be diagnosed with the use of ANN without undergoing a sleep study, and that empiric management with auto-CPAP has similar outcomes to those who undergo a formal sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult (≥18 years old)
* Must have symptoms suggestive of OSA, and be considered for sleep study by the sleep specialist provider.

Exclusion Criteria:

* Pregnancy or breast feeding
* Patients with severe congestive heart failure (eg, NYHA Class IV, ejection fraction < 35%).
* Patients with end-stage renal disease on hemodialysis
* Patients with CVA, Parkinson, neuromuscular degenerative disease.
* Patient on narcotics.
* Patients with severe lung disease requiring oxygen at night and/or during the day.
* Patient with predominant insomnia or sleep hygiene problems, and who are not considered for PSG by the sleep specialist.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate that using an ANN directed management of OSA is not inferior to PSG directed management of OSA in terms of sleepiness related functional outcome | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ali El-Solh, MD, MPH, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Veterans Affairs Medical Center in Buffalo, Buffalo, New York, United States